CLINICAL TRIAL: NCT01586858
Title: Rituximab for Anti-neutrophil Cytoplasmic Antibodies (ANCA)-Associated Vasculitis (RAVE) Long-Term Follow-Up Study
Brief Title: Rituximab for ANCA-associated Vasculitis (RAVE) Long-Term Follow-Up Study
Acronym: RAVELOS
Status: Terminated | Type: Observational
Why Stopped: Loss of Funding
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Alabama at Birmingham (Other); Boston University (Other); Mayo Clinic (Other); Duke University (Other); The Cleveland Clinic (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: ML27815
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Granulomatosis With Polyangiitis; Microscopic Polyangiitis
Keywords: Vasculitis; ANCA; Rituximab; Small vessel vasculitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Vasculitis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RAVE subjects
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational study of subjects previously enrolled in the RAVE trial

SUMMARY:
Rituximab is the first drug approved by the United States Food and Drug Administration (FDA) for the treatment of patients with granulomatosis with polyangiitis (Wegener's granulomatosis) or microscopic polyangiitis. Because it is a relatively new medication, the long-term safety and efficacy of this drug is not yet clear. This study proposes to follow patients who were enrolled in the RAVE study to determine if treatment with rituximab influences long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in the RAVE trial
2. Completion of RAVE Common Closeout Date visit
3. Informed consent

Exclusion Criteria:

1. Refusal to participate
2. Inability to comply with standard-of-care, including routine clinical visits and testing.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RAVE study participants
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-05-15 (Actual); Study Completion 2014-05-15 (Actual)

PRIMARY OUTCOMES:
Long-term safety of rituximab for the treatment of ANCA-associated vasculitis | Four years
  To determine the long-term safety of rituximab for the treatment of ANCA-associated vasculitis (granulomatosis with polyangiitis (Wegener's granulomatosis) and microscopic polyangiitis).

SECONDARY OUTCOMES:
Disease activity | Four years
  Disease activity, assessed by the proportion of patients with severe flares
Disease damage assessed by the increase in Vasculitis Damage Index (VDI) | Four years
  The VDI is composed of 11 categories (e.g., musculoskeletal, pulmonary) and 64 individual damage items. The score ranges from 0 (no damage) to 64 (all individual damage items).
Disease damage assessed by the ANCA-Vasculitis Index of Damage (AVID) | Four years
  The AVID has 12 categories and 112 individual damage items. The score ranges from 0 (no damage) to 129 (all individual damage items). Although there are 112 items, 17 items are related to eyes and ears and can be scored for left, right or both.
Renal survival | Four years
  Renal survival, assessed by the proportion of patients doubling their serum creatinine, reaching Stage V Chronic Kidney Disease (defined as a glomerular filtration rate ≤15 ml/min), or both.
Malignancy | Four years
  Proportion of patients with incident malignancies, including type of malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Philip Seo, MD, Study Director — Johns Hopkins University
Locations (8):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Mayo Clinic Foundation, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Duke University, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
- University Hospital Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199